CLINICAL TRIAL: NCT03826394
Title: The Effects of Exercise and Dietary Interventions in Overweight and Obese Postpartum Women on Weight Management and Health.
Brief Title: Lifestyle Interventions in Overweight and Obese Postpartum Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nottingham Trent University (Other)
Responsible Party: Principal Investigator, Stephanie Hanley, Miss, Nottingham Trent University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NottinghamTU
Record Dates: First submitted 2019-01-28; First posted 2019-02-01 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Overweight and Obesity
Keywords: Postpartum, Overweight, Obesity, Exercise, Diet, Lifestyle
MeSH Terms: conditions — Overweight; Obesity; Motor Activity | interventions — Diet Therapy

STUDY DESIGN:
Intervention Model Description: Participants will take part in an exercise or dietary intervention in a non-randomised, parallel study.
  Each intervention will be preceded by a four week tracked free-living period. Both interventions will be completed over a sixteen week period. Following the tracked period, participants will choose to take part in either the exercise or dietary intervention. Intervention information will be delivered in four, three week blocks. No new information will be provided during the final four weeks of the intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Intervention (Experimental): Exercise intervention with the aim of incrementally increasing physical activity to meet the national recommendation of 150 minutes a week of moderate-vigorous physical activity, reducing BMI and improving overall health.
  Interventions: Behavioral: Exercise Intervention
- Dietary Intervention (Experimental): Staged dietary intervention with the aim of improving eating behaviours, reducing BMI and improving overall health.
  Interventions: Behavioral: Dietary Intervention

INTERVENTIONS:
Behavioral: Exercise Intervention — Education based sixteen week intervention where participants will be provided with core information every three weeks and supplementary information through technological means at other time points. All provided information will be exercise specific. Individualised and group support provided throughout the first twelve weeks and withdrawn for the final four weeks. Fitbit Flex 2 provided for the duration of the study.
  Other Names: Physical Activity Intervention
  Arms: Exercise Intervention
Behavioral: Dietary Intervention — Education based sixteen week intervention where participants will be provided with core information every three weeks and supplementary information through technological means at other time points. All provided information will be diet specific. Individualised and group support provided throughout the first twelve weeks and withdrawn for the final four weeks. Fitbit Flex 2 provided for the duration of the study.
  Other Names: Nutritional Intervention/Healthy eating Intervention
  Arms: Dietary Intervention

SUMMARY:
The current study aims to investigate the effects of a chosen technology-based exercise or healthy eating intervention that combines individual and group-based support, on weight loss and other health-related parameters in postpartum women with overweight or obesity. All participants will be asked to engage in a 20-week programme consisting of a 4 week tracked free living period followed by a 16-week intervention. The investigators hypothesise that reductions in BMI (body mass index) and improvements in health-related parameters will be observed post-intervention.

DETAILED DESCRIPTION:
The current study will investigate the effects of a chosen exercise or dietary intervention on BMI and other health-related parameters in postpartum women with overweight and obesity. Dietary or physical activity interventions, alone or combined, are associated with greater weight loss when provided to women in the postpartum period, compared with no intervention. Providing a combined physical activity and dietary intervention is associated with an average weight loss of 2.49kg post-intervention and 2.4kg 12 months after pregnancy. However, the variation in average weight loss achieved is great which could be due to differences in the design of lifestyle programmes.

Interventions including individualised support and self-monitoring have proven more effective in promoting reductions in BMI in postpartum women. However, high levels of attrition and poor engagement have been highlighted as two areas that require attention in this area. Therefore, future research is required to identify strategies best suited to the design and implementation of effective lifestyle interventions in overweight and obese postpartum women.

Women between six weeks and one year postpartum will elect to be part of either a 16-week exercise or dietary intervention. Prior to this, participants will be tracked for a period of four weeks in free living conditions. Each intervention will be split into four blocks of three weeks where staged intervention specific information will be provided. Individualised face-to-face and technological group support will be provided throughout. For the final four weeks of the intervention no new information will be provided and all support will be withdrawn.

Analyses of body composition and girths, blood metabolites, resting heart rate, blood pressure, and questionnaires assessing physical activity, eating behaviours and quality of life will be carried out alongside assessments of BMI at baseline, pre-intervention and at both twelve and sixteen weeks of the intervention. Measures of BMI, resting heart rate, blood pressure and questionnaire scores will be taken at each three weekly stage of the intervention.

ELIGIBILITY:
Inclusion Criteria:

Be at least 18 years old at the date of their first visit. Have a body mass index (BMI) of greater than 25 kg∙m2 (this will be worked out by the researchers using the participant's height and body weight). Have had a singleton pregnancy. Have had one pregnancy to date. Be 6 weeks-1 year postpartum (and had physician's approval to return to exercise).

Own a smartphone (able to download and use WhatsApp). In the researcher's opinion, the participant is able and willing to follow all trial requirements.

Exclusion Criteria:

Have a clinical diagnosis of depression/postnatal depression. Currently enrolled on another weight loss programme. Currently consuming weight loss tablets/supplements. Have heart/liver/chronic renal disease. Have a clinical diagnosis of Type 2 Diabetes Mellitus. Consume excessive amounts of alcohol (regularly drinking more than 14 units of alcohol a week). Actively trying for another baby/planning a pregnancy in the next 6 months. Experienced a stillbirth. Have any health conditions that affect physical activity engagement. On any medication that affects the ability to exercise. On any medication that affects the ability to follow a healthy eating programme.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2019-08-19 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Changes in BMI | Week 0, 4, 7, 10, 13, 16, 20
  Weight (kg) and height (m) will be combined to report BMI in kg/m^2

SECONDARY OUTCOMES:
Change in Body Composition | Week 0, 4, 16, 20
  Whole body DXA (dual energy X-ray absorptiometry) scan to assess fat mass, fat-free mass, bone density.
Change in Blood Metabolites | Week 0, 4, 16, 20
  Fingertip blood sample taken to assess total cholesterol, high-density lipoprotein cholesterol, low-density lipoprotein cholesterol, triglycerides, glycated haemoglobin, random glucose.
Change in Body Girths | Week 0, 4, 16, 20
  Measures (in cm) of waist, hip, thigh, calf, bust and upper arm girths.
Change in Blood Pressure | Week 0, 4, 7, 10, 13, 16, 20
  Measure of blood pressure taken at rest.
Change in Resting Heart Rate | Week 0, 4, 7, 10, 13, 16, 20
  Measure of heart rate taken at rest.
Change in Quality of Life | Week 0, 4, 7, 10, 13, 16, 20
  Assessment of quality of life using the Impact of Weight on Quality on Life (Lite) and Short-Form 36 Questionnaires.
  Short-Form 36- scores range from 0-100 (lower scores= more disability; higher scores = less disability).
  Impact of Weight on Quality of Life- 31-item that calculates a total score and scores on 5 separate domains (physical function, self-esteem, sexual life, public distress, work).
Change in Sleep Quality | Week 0, 4, 7, 10, 13, 16, 20
  Assessment of sleep quality using Pittsburgh Sleep Quality Index Questionnaire. Index contains 19 self-rated questions and 5 questions rated by the bed partner or roommate. Only self-rated questions are included in the scoring. Self-rated items are combined to form 7 component scores, each of which has a range of 0-3 points. A score of 0 indicates no difficulty while a score of 3 indicates severe difficulty. The 7 components scores are then summed together to yield one global score, with a range of 0-21 points. 0 indicates no difficulty and 21 indicates severe difficulties in all areas.
Change in Eating Behaviours | Week 0, 4, 7, 10, 13, 16, 20
  Assessment of eating behaviours using Three Factor Eating Questionnaire. Responses to each of the 18 items are given a score of between 1 and 4 and item scores are summated into scale scores for cognitive restraint, uncontrolled eating and emotional eating. Higher scores in the respective scales are indicative of greater cognitive restraint, uncontrolled, or emotional eating.
Change in Physical Activity Levels | Week 0, 4, 7, 10, 13, 16, 20
  Measures of physical activity levels through direct (Fitbit) and indirect (Godin 7-day leisure time physical activity questionnaire) measures.
Change in Markers of Postnatal Depression | Week 0, 4, 7, 10, 13, 16, 20
  Assessment of markers of depression using Edinburgh Postnatal Depression Scale. Responses to each of the 10 items are given a score of 0 to 3. The maximum score is 30. Higher scores indicate greater degrees of depression, with a score of 13 or above indicating varying degrees of depressive illness.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie J Hanley, MRes, Principal Investigator — Nottingham Trent University
Locations (1):
- Nottingham Trent University, Clifton Campus, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data may be made available to other researchers following completion of the current trial in an anonymised/pseudonymised format to prevent individual participant identification. Data will be provided in response to certain requests (e.g. if a systematic review and meta-analysis/statistical power calculation is being conducted that requires access to certain raw data).

REFERENCES:
- [Background] McKinley MC, Allen-Walker V, McGirr C, Rooney C, Woodside JV. Weight loss after pregnancy: challenges and opportunities. Nutr Res Rev. 2018 Dec;31(2):225-238. doi: 10.1017/S0954422418000070. Epub 2018 Jul 9. PMID 29984681
- [Background] Dalrymple KV, Flynn AC, Relph SA, O'Keeffe M, Poston L. Lifestyle Interventions in Overweight and Obese Pregnant or Postpartum Women for Postpartum Weight Management: A Systematic Review of the Literature. Nutrients. 2018 Nov 7;10(11):1704. doi: 10.3390/nu10111704. PMID 30405088
- [Background] Dodd JM, Deussen AR, O'Brien CM, Schoenaker DAJM, Poprzeczny A, Gordon A, Phelan S. Targeting the postpartum period to promote weight loss: a systematic review and meta-analysis. Nutr Rev. 2018 Aug 1;76(8):639-654. doi: 10.1093/nutrit/nuy024. PMID 29889259
- [Background] Guo J, Chen JL, Whittemore R, Whitaker E. Postpartum Lifestyle Interventions to Prevent Type 2 Diabetes Among Women with History of Gestational Diabetes: A Systematic Review of Randomized Clinical Trials. J Womens Health (Larchmt). 2016 Jan;25(1):38-49. doi: 10.1089/jwh.2015.5262. Epub 2015 Dec 24. PMID 26700931
- [Background] Burke LE, Wang J, Sevick MA. Self-monitoring in weight loss: a systematic review of the literature. J Am Diet Assoc. 2011 Jan;111(1):92-102. doi: 10.1016/j.jada.2010.10.008. PMID 21185970